CLINICAL TRIAL: NCT07293858
Title: Optical Coherence Tomography: Prognostic Value and Artificial Intelligence
Acronym: ORANGE
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-13271
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Arterial Disease
Keywords: Optical Coherence Tomography; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the prognostic value of optical coherence tomography (OCT) imaging of the coronary arteries. OCT provides high-resolution images of the vessel wall and stented segments during routine cardiac catheterization. All patients who undergo OCT as part of their clinical care are invited to participate in this prospective registry.

The study will examine whether specific OCT-derived characteristics-such as plaque morphology, vulnerable features, or indicators of stent optimization-are associated with long-term clinical outcomes. Follow-up information on symptoms, medication use, hospitalizations, cardiac procedures, and major cardiac events will be collected through medical records, questionnaires, and national registry data over a period of up to 10 years.

In addition, pseudonymized OCT pullbacks will be used to support the development of an artificial intelligence (AI) algorithm for automated annotation of OCT images. This algorithm may help improve the clinical interpretation of OCT by identifying relevant imaging features in a consistent and efficient manner.

Participation is voluntary and includes permission to use clinical data, OCT images, and follow-up information for research purposes. Data are coded to protect participant privacy and stored securely according to applicable regulations. The results of this study may contribute to better understanding of coronary plaque characteristics and may support improved decision-making in interventional cardiology.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing intracoronary OCT imaging at the Radboud University Medical Center, and any additional centers that may join the study in the future.
* OCT performed at the discretion of the treating physician, according to contemporary clinical guidelines.
* Written informed consent obtained after the procedure.

Exclusion Criteria:

* Patients who decline or are unable to provide informed consent. (Only patients who provide consent can be included.
* Patients for whom follow-up or data collection is not feasible (e.g., no valid contact details).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all patients who have undergone intracoronary OCT imaging of the coronary arteries as part of their routine cardiac catheterization. This is an all-comer population with no restrictions regarding indication, diagnosis, age, or comorbidities. The decision to perform OCT is made independently by the treating cardiologist. After the procedure, patients are invited to participate in this prospective registry and are included only after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between OCT-derived plaque and stent characteristics and long-term clinical outcomes | 10 years
  Assessment of whether specific OCT-derived characteristics-such as plaque morphology, vulnerable features, stent deployment quality, and other intraluminal or vessel wall findings-are associated with long-term clinical outcomes. Outcomes include cardiac symptoms, cardiac events, coronary interventions, hospitalization, and death, based on medical records, questionnaire data, and national registries.

SECONDARY OUTCOMES:
Performance of an automated OCT annotation algorithm | Baseline (OCT acquisition) to algorithm development period (≤5 years)
  Evaluation of the accuracy and feasibility of an AI-based algorithm for automated annotation of OCT pullbacks. Pseudonymized OCT images will be used to train and validate automated detection of plaque features, stent characteristics, and other relevant imaging markers. Comparison will be made with expert manual annotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands